CLINICAL TRIAL: NCT01084720
Title: Efficacy, Local Tolerance and Patient Acceptability of a Moisturizing Emollient in Patients Undergoing Maintenance Renal Dialysis With Uremic Xerosis (MRD)
Brief Title: Efficacy, Local Tolerance and Patient Acceptability of a Moisturizing Emollient in Patients With Uremic Xerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Orfagen (Industry)
Responsible Party: Dr Patrick Dupuy, MD, Orfagen
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: V00034 CR 302 (ORF)
Record Dates: First submitted 2010-03-09; First posted 2010-03-10 (Estimated); Last update posted 2010-03-10 (Estimated); Status verified 2010-03

CONDITIONS: Uremic Xerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: V0034 CR

SUMMARY:
* To evaluate the palliative effects of a moisturising emollient, in patients with uremic xerosis of moderate, severe or very severe intensity, associated or not to uremic pruritus.
* To assess the local tolerance of the test product and its vehicle, and to evaluate the overall agreement (efficacy, tolerance easiness of use) of the patients for the test product.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes, of at least 10 years of age
* Patients undergoing either hemodialysis or peritoneal dialysis due to chronic renal failure
* Patients whose xerosis is related to their renal insufficiency status
* Patients suffering from moderate to severe xerosis, i.e. with a severity score of at least 2, on two symmetric areas of the lower legs (Phase I test areas)
* Patients who have not experienced phototherapy within 8 weeks prior to study entry
* Patients with no antipruritic treatment, or with stable antipruritic treatments (e.g. antihistamines, cholestyramine, opioid inhibitors, charcoal) at least 4 weeks before study entry
* Written informed consent (Appendix II) from the patients or parents

Exclusion Criteria:

* Patients under 10 years of age
* Patients undergoing renal dialysis for another reason than MRD
* Patients whose xerosis or pruritus is due to another reason than their MRD status
* Patients suffering from mild xerosis (score £ 1) on the lower legs
* Patients with xerosis of non comparable severity between the lower legs
* Patients with a known history of allergy to one of the ingredients contained in the test product
* Patient with an intercurrent condition which may interfere with a good conduct or the study parameters of the study
* Patients treated with any other emollient/moisturizing topical preparation within the 7 days prior to study entry
* Patients with phototherapy within 8 weeks prior to study entry
* Patients who started an antipruritic treatment other than phototherapy, or who experienced unstable dosage schedule of antipruritic treatments (e.g. antihistamines, cholestyramin, opiod inhibitors, charcoal) within 4 weeks prior to study entry
* Patients who participated in a study within the 3 months prior to study entry
* Patients who are not able or willing to follow the study instructions
* Patients or parents who refuse to give written informed consent

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2002-12; Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Severity of uremic xerosis on the lower legs on day 7 | 7 days
  Severity of uremic xerosis on the lower legs on day 7 by the investigator, using a defined 5-point severity scale. A therapeutic response was defined as a decrease of at least 2 grades of the xerosis after 7 days (end of phase I).

SECONDARY OUTCOMES:
Local tolerance of the test product and its vehicle and overall agreement (efficacy, tolerance easiness of use) of the patients for the test product. | 56 days

CONTACTS AND LOCATIONS:
Overall Officials: Jacek Szepietowski, Professor, Principal Investigator — DEPT. OF DERMATOLOGY, UNIVERSITY OF MEDICINE, UL. CHALUBINSKIEGO, POLAND